CLINICAL TRIAL: NCT02961387
Title: A Clinical Trial on Effectiveness and Safety of Inhaling Hydrogen-oxygen to Decreases Inspiratory Effort for the Patients With Tracheal Stenosis: A Randomized, Double-blind and Single-center Clinical Study
Brief Title: A Clinical Trial on Effectiveness and Safety of Hydrogen Generator to Treat Dyspnea for the Patients With Tracheal Stenosis: A Randomized, Double-blind and Single-center Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Professor of Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TS20160801
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Tracheal Stenosis
Keywords: Tracheal stenosis, Hydrogen generator, Hydrogen-oxygen, Dyspnea.
MeSH Terms: conditions — Tracheal Stenosis; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrogen generator treatment (Experimental): Inhalation of hydrogen-oxygen mixed gas.
  Interventions: Device: Hydrogen generator treatment; Device: Oxygen-making machine treatment
- Oxygen-making machine treatment (Sham Comparator): Inhalation of oxygen.
  Interventions: Device: Hydrogen generator treatment; Device: Oxygen-making machine treatment

INTERVENTIONS:
Device: Hydrogen generator treatment — The patients mainly used the hydrogen generator with nebulizer for inhalation of hydrogen-oxygen mixed gas.
Device: Oxygen-making machine treatment — The patients mainly used medical molecular sieve oxygen-making machine for oxygen inhalation.

SUMMARY:
Investigators aim to study the effectiveness and safety of inhaling hydrogen-oxygen which produced by a hydrogen generator with nebulizer to decreases inspiratory effort for the patients with tracheal stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 65;
2. Diagnosed moderate/severe tracheal stenosis by chest CT and/or bronchoscopy;
3. Difficulty breathing symptoms
4. Agree to participate in this trial and sign the informed consent form.

Exclusion Criteria:

1. Those who were suffered from respiratory failure or more severe caused by dyspnea;
2. Combined other serious systemic diseases (severe arrhythmia, acute myocardial ischemia, uncontrollable hypertension crisis, active gastric ulcer, uncontrolled diabetes, renal failure, blood system diseases or coagulation dysfunction);
3. Those who were suffered from severe mental illness or could not take care of themselves;
4. Pregnant or lactating women;
5. Those who could not understand the trial procedures and correctly the trial equipment;
6. Those who participated in other clinical trials in the first 3 months before the screening date.

Quit criteria

1. The subjects requiring emergency intubation or other intervention or surgical treatment due to worsened tracheal stenosis;
2. Subjects who had severe adverse events during treatment;
3. Subjects who did not want to continue to participate in the trial;
4. The subjects who were necessarily terminated for the trial by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in sRMSdi/para/sc, RMSdi, Pdi& MIP from baseline after inhalation by bench study. | Baseline, 10min, 20min, 30min, 40min, 50min, 90min and 150min
  sRMSdi/para/sc: root-mean-square of diaphragm/parasternal/sternocleidomastoid surface electromyography; RMSdi: root-mean-square of diaphragm electromyography; Pdi: Transdiaphragmatic pressure; MIP:maximal inspiratory pressure.

SECONDARY OUTCOMES:
Change in Borg score for dyspnea after inhalation. | Baseline, 10min, 20min, 30min, 40min, 50min, 90min and 150min
Change in symptom of dyspnea from baseline after inhalation. | Baseline, 10min, 20min, 30min, 40min, 50min, 90min and 150min
  Changes in comfort with each gas mixture were evaluated by a simple questionnaire
Change in signs(BR, HR, BP, el) from baseline after inhalation | Baseline, 10min, 20min, 30min, 40min, 50min, 90min and 150min
  Change in signs include breath rate， heart rate， blood pressure，Three Depression Sign and so on.
Change in PaO2, PaCO2, PH& HCO3- after inhalation | Baseline and 150min
  Change in Arterial blood gases.
FEV1 & FVC | Baseline
  Forced expiratory volume in one second & Forced vital capacity.
Change in impulse oscillometry variables(R5,R20,X5,AX,RF) as change from baseline when inhaling. | Baseline and inhaling
  R5 - Resistance at 5Hz, R20 - Resistance at 20Hz, X5 - Reactance at 5Hz, RF - Frequency of resonance, AX - Area under reactance curve
Change in cough waves from baseline when inhaling | Baseline, Inhaling.
  Cough waves will be recorded by a voice recorder.
Grades of airway stenosis by bronchoscopy | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China